CLINICAL TRIAL: NCT05049291
Title: Pilot Study of an Advance Care Planning Intervention Among Persons With Dementia in Long-term Services and Support Facilities
Brief Title: Pilot Study of an Advance Care Planning Intervention Among Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Donald Sullivan, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00021951
Record Dates: First submitted 2021-08-25; First posted 2021-09-20 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Advanced Care Planning; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): One time receipt and review of an information sheet
  Interventions: Behavioral: telehealth advance care planning
- Non-Intervention (No Intervention): Usual care will be delivered per standards of care.

INTERVENTIONS:
Behavioral: telehealth advance care planning — An education information sheet containing prognosis and outcomes of acute care and intensive treatments
  Arms: Intervention

SUMMARY:
Advance care planning allows people to have their wishes taken into account even in the advanced stages of the persons' condition and at the end of life when the person may be unable to communicate. However, a recent review found an absence of high-quality guidelines for advanced care planning in dementia care. Since few evidence-based resources exist, the investigators propose a study to generate, refine, and pilot test an education information sheet designed to promote advanced care planning among families of persons with dementia.

DETAILED DESCRIPTION:
To determine the feasibility, acceptability and preliminary efficacy of an education information sheet to promote advance care planning among family members of persons with advanced dementia in long-term services and support facilities.

Introducing an education information sheet containing prognosis and outcomes will be feasible, acceptable, and increase self-efficacy and do-not-hospitalize decision preferences among family members of persons with advanced dementia.

ELIGIBILITY:
Inclusion Criteria:

* Family member of a person with a diagnosis of dementia (any type)
* English-speaking family member
* Family member of a person with dementia admitted to a nursing home

Exclusion Criteria:

* Inability to understand/read English
* Advance directive already in patient chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of Information Sheet among Study Population | 6 months
  Feasibility of the information sheet is defined as the consent rate of family members who are offered enrollment. This will be calculatd as a percent of family members (number of enrolled participants/number of eligible participants offered enrollment)
Acceptibility of Decision Aid Tool | 6 months
  Acceptability using an adapted tool (https://decisionaid.ohri.ca/eval_accept.html) which measures the ratings of comprehensibility of the information sheet among participants in the intervention group. Responses are reported descriptively in terms of proportions responding positively or negatively on each criteria.

SECONDARY OUTCOMES:
Decision Self-efficacy Scale | 6 months
  Measures self-confidence or belief in one's abilities in decision making, including shared decision making. Eleven responses are measured on a 0-4 likert scale and a final summed scale is converted to a 0-100 range (scores are summed, divided by 11, then multiplied by 25). A score of zero means low self efficacy and score of 100 means extremely high self efficacy.
Family Member Decision-Making Self-Efficacy Scale | 6 months
  Measures family member self-efficacy in medical decision-making on behalf of a loved one. This scale has two versions, one for conscious and one for unconscious loved ones, which we will use accordingly. Thirteen items are measured on a 0-5 Likert scale with 1 being "cannot do at all" and 5 being "certain I can do." Higher scores indicate higher decision making self-efficacy.
Adaptation of Advance Care Planning Engagement Survey | 6 months
  Questions adapted from an 82-item questionnaire that measures advance care planning engagement in terms of knowledge, contemplation, self-efficacy and readiness. We include 10 questions from the measure. We used a mean imputation approach. All available data were included to create an average 5-point Likert score.
Preparation for Decision-Making Scale | 6 months
  Measures perception of the usefulness of a decision support tool in preparing respondent for decision-making. Responses are on a Likert scale of 1-5 with one being "not at all" and five being " a great deal." Items are summed for scoring. A higher score indicates a higher level of perceived helpfulness in preparing for decision-making.
Adaptation of Advance Care Planning Engagement for Surrogates Survey | 6 months
  We adapted 9 items from the 17-item Advance Care Planning for Surrogates survey. Response options are on a 5-point Likert scale. We will calculate a summary score, with higher scores indicates a higher level of engagement.
Knowledge about Dementia | 6 months
  Six questions to assess family members' knowledge about dementia were developed for this pilot study. All questions are true/false. Each correct answer will be coded as 1, each incorrect answer will be scored as 0. Higher scores indicate more knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States